CLINICAL TRIAL: NCT00944736
Title: Effect of Probiotic VSL#3 on Intestinal Permeability of Pediatric Patients With Crohn's Disease in Remission
Brief Title: Effect of VSL#3 on Intestinal Permeability in Pediatric Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: VSL Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Julia Bracken, Assistant Professor of Medicine, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09 06-115
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Pediatric; VSL#3; Permeability; Probiotic; Zonulin
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSL#3 (Active Comparator)
  Interventions: Dietary Supplement: VSL#3
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — 1 packet BID
  Arms: VSL#3
Dietary Supplement: Placebo — 1 inactive packet BID
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of a probiotic formulation, VSL#3, on intestinal permeability in pediatric patients with Crohn's disease.

DETAILED DESCRIPTION:
Children with Crohn's disease have altered intestinal permeability. A pilot study in children showed that probiotics may decrease intestinal permeability. In this double blind, randomized controlled trial, we will observe the effect of VSL#3 on small bowel permeability using a double sugar absorption test. PCDAI was monitored, but not analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of small bowel or colonic Crohn's disease as defined by histological and endoscopic criteria.
* Males or females ages 11-17 years.
* Crohn's disease in remission as defined by a Pediatric Crohn's Disease Activity Index (PCDAI) < 10
* Patients on maintenance doses of aminosalicylates, 6-MP and/or Azathioprine for at least 2 months.
* Procurement of written informed consent signed by the subject's legal guardian and study investigator(s) and patient assent.

Exclusion Criteria:

* Patients with documented intestinal stricture.
* Patients with signs of symptoms of systemic or intestinal infection.
* Antibiotic use the previous 1 month.
* Probiotic use in the previous 2 months (excluding yogurt).
* Use of the following medications; Methotrexate, Cyclosporine, Tacrolimus and Infliximab.
* Patients with diagnosis of other co-morbid diseases such as heart disease, renal disease, immunodeficiency, diabetes, or thyroid disease.
* Patients with indwelling catheters.
* Patients with short bowel syndrome
* Positive urine pregnancy test for female subjects

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Intestinal Permeability - measured by Sugar Absorption Test | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia M Bracken, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States